CLINICAL TRIAL: NCT02291224
Title: Development and Testing of a Clinic-Based Intervention to Increase Dual Protection Against Unintended Pregnancy and Sexually Transmitted Diseases (STDs) Among High Risk Female Teens
Acronym: 2Gether
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Emory University (Other); Grady Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-6588; DP12-001 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2014-07-24; First posted 2014-11-14 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy; Sexually Transmitted Diseases
Keywords: dual protection; pregnancy; reproductive health; sexually transmitted diseases; condoms; contraception; adolescent health services
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Other): The control arm receives the clinic standard of care counseling. This includes individual clinical care and counseling consistent with protocols at the Grady Health System Teen Services Clinic, with study visits at enrollment, 6 months, and 12 months, during which any medical care or counseling included in the clinic standard of care will be provided. All control group members will see a provider on the day of enrollment. Control arm participants will get phone calls from clinic staff to update their contact information and remind them of upcoming appointments at 3 weeks and 5 months after both the enrollment visit and the 6 month visit. Participants may visit the clinic at any time and will be encouraged to come into the clinic for any concerns. If they have an interim visit during the study period, they will receive the clinic standard of care.
  Interventions: Behavioral: Standard of care counseling
- Intervention (Experimental): 1. Enrollment
     * Interactive multimedia platform focused on DP strategies.
     * Intervention arm counseling by a health care provider to select DP strategy.
     * Intervention arm counseling and skill-building by a nurse educator (NE) on correct, consistent use of DP strategy.
  2. Booster counseling by an NE via phone at 3 weeks and 5 months after both the enrollment visit and the 6 month visit.
  3. 6 month visit
     * Abbreviated version of the interactive multimedia platform on DP strategies and adherence.
     * Intervention arm counseling by an NE to reinforce skills for correct, consistent use of DP strategy.
  4. Interim visits: Participants may visit the clinic at any time. If intervention group members visit the clinic for STI treatment or to switch birth control method, providers and/or NEs will follow structured counseling guides. If they have an interim visit for another reason, they will receive the clinic standard of care.
  Interventions: Behavioral: Interactive multimedia platform; Behavioral: Intervention arm counseling

INTERVENTIONS:
Behavioral: Interactive multimedia platform — An interactive platform that includes video vignettes of young women who are choosing dual protection strategies (based on a synthesis of focus group data from members of the TSC patient population), as well as true/false questions to build knowledge about dual protection and dispel common myths about contraceptive strategies. There will also be reflection questions that encourage participants to consider values and priorities in their own lives that may influence their dual protection strategy selection.
  Other Names: MMDP
  Arms: Intervention
Behavioral: Intervention arm counseling — Counseling for the intervention group will follow carefully developed guides and incorporate the participants' answers to the reflection questions in the interactive multi-media component. This counseling has a set structure (set forth in separate counseling guides for health care providers and nurse educators), incorporates motivational interviewing techniques, includes multiple opportunities for role play, and is designed to be patient-centered.
  Arms: Intervention
Behavioral: Standard of care counseling — Standard of care counseling is provided by health care providers and health educators at TSC. It incorporates extensive counseling on methods to prevent both unintended pregnancy and sexually transmitted infections, however the structure of the counseling and techniques used are dependent on the standard practice of each provider or educator. This counseling does not incorporate answers to reflection questions from the multi-media platform because control arm participants will not view this content.
  Arms: Control

SUMMARY:
This trial will evaluate a multi-component, clinic-based intervention aimed at increasing dual protection strategy selection and adherence among young African American females at an urban family planning clinic. Dual protection is the use of contraceptive strategies to prevent both unintended pregnancy (UIP) and sexually transmitted infections (STIs). This is an unblinded randomized controlled trial; participants will either get the interactive multimedia platform focused on DP strategies with intervention arm counseling or the standard of care arm counseling.

The study will recruit 710 African American females aged 14-19 who are attending the Grady Health System (GHS) Teen Services Clinic (TSC) in Atlanta, Georgia, for reproductive health care.

The trial will recruit and enroll 710 young women presenting to the clinic for clinical care who have the following characteristics:

* self-identify as African American,
* 14-19 years of age,
* have had vaginal sex with a male partner in the past 6 months,
* HIV-negative by self-report,
* not pregnant,verified by urine pregnancy test,
* no desire to be pregnant in next 12 months,
* plan to stay in the Atlanta area for the next year,
* are willing to provide contact information, and
* were not previously enrolled in the pilot study of this intervention.

Those enrolled will be in the study for 12 months. Young women who are eligible and give written consent or assent for study participation will be enrolled. Half will be randomized to the control arm, half to the intervention arm.

1. Control arm (standard of care) includes individual clinical care and standard of care counseling consistent with protocols at the TSC, with study visits for data collection at enrollment, 6 months, and 12 months, during which any medical care or counseling that they would normally get will also be provided. Control arm participants will also get telephone calls from clinic staff to update their contact information and remind them of upcoming visits at 3 weeks and 5 months after the enrollment visit, and at 3 weeks and 5 months after the 6 month visit.
2. Intervention arm, consisting of the following intervention components:

   1. Enrollment visit

      * A culturally-appropriate interactive multimedia platform focused on DP strategies and designed to prepare the individual for selection of a DP strategy.
      * Individual intervention arm counseling to select the DP strategy that is best suited for the participant (by a clinic health care provider).
      * Individual intervention arm counseling to build skills for correct and consistent use of the selected DP strategy (by a nurse educator (NE)).
   2. Booster counseling via phone at about 3 weeks and 5 months after the enrollment visit, and at about 3 weeks and 5 months after the 6 month visit (by an NE).
   3. 6 month visit

      * An abbreviated version of the interactive multimedia platform focused on dual protection strategies and strategy adherence.
      * Individual intervention arm counseling to reinforce skills for correct and consistent use of the DP strategy (by an NE).

At the final study visit at 12 months there is no difference between the counseling provided to the two groups; participants in both arms will receive the clinic standard of care.

Participants in both arms of the study will follow the same data collection procedures throughout the study:

* At all three study visits, participants in both arms will receive urine pregnancy and STI tests and complete an audio computer assisted self-interview (ACASI) questionnaire.
* At 3 and 9 months after enrollment, participants in both arms will receive a data collection call with administration of a telephone questionnaire.

Throughout the study, all participants will be encouraged to come in for evaluation if they have any concerns. Any data from pregnancy or STI testing at these interim clinic visits will be later collected via chart review. If participants seek reproductive health care at other facilities during the study period, records will be requested with participant permission, and data from pregnancy or STI testing at these outside clinic visits will be collected via review of records received.

We will examine the efficacy of the intervention arm relative to control arm across the following primary behavioral and biologic outcomes over the 12 months of follow-up:

1. Self-reported dual protection strategy selection
2. Self-reported dual protection strategy adherence
3. Incidence of pregnancy or infection with chlamydia, gonorrhea or trichomonas (as confirmed by laboratory testing)

A small pilot study was be conducted prior to the initiation of enrollment in the main study.

ELIGIBILITY:
Inclusion Criteria:

* female,
* self-identify as African American,
* 14-19 years of age,
* present to clinic on date of potential enrollment for clinical care,
* has had vaginal sex with a male partner at least once in the past 6 months,
* HIV-negative by self-report,
* not currently pregnant (verified by urine pregnancy test),
* desire to avoid pregnancy for at least 12 months,
* plan to be in the Atlanta area for the next 12 months,
* competent to participate in consenting or assenting process per recruiter evaluation,
* willing to provide contact information, and
* not previously enrolled in the pilot study of this intervention.

Exclusion Criteria:

* pregnant
* HIV positive

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 709 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Participant selection of an effective dual protection (DP) strategy | 6 months
  Whether or not a participant self-reports having selected an effective DP strategy. An effective DP strategy is defined as one of the following:
  * Abstinence from vaginal sex;
  * Effective non-barrier contraceptive method [including intrauterine device (IUD), Implant, Depo, or contraceptive pill, patch or ring] with consistent condom use;
  * Consistent condom use only
Participant report of adherence to DP strategy | 3 months
  By self-report from audio computer-assisted self-interviewing (ACASI) and telephone questionnaires; adherence is measured by three different outcomes:
  * Whether or not DP strategy was used at last sex
  * Whether or not DP strategy was used consistently during last 3 month time period
  * Estimated proportion of time adherent to DP strategy over last 3 months
Time to first biologic event (pregnancy or diagnosis with STI) in participants | Within 12 month period following enrollment
  Measured by date of positive lab test ("biologic event" refers to a positive pregnancy test or diagnosis with chlamydia, gonorrhea or trichomonas infection).
Incidence of pregnancy and sexually transmitted infections (STIs) | Within 12 month period following enrollment
  Includes the proportion of participants with a lab-confirmed diagnosis of pregnancy or lab-confirmed diagnosis with infection with chlamydia, gonorrhea or trichomonas within the 12 month follow-up period (testing either performed at study site clinic and documented at study visits and via chart review, or diagnosed by outside labs with documentation obtained via release of information procedures)
Participant selection of an effective dual protection (DP) strategy | 12 months
  Whether or not a participant self-reports having selected an effective DP strategy. An effective DP strategy is defined as one of the following:
  * Abstinence from vaginal sex;
  * Effective non-barrier contraceptive method [including intrauterine device (IUD), Implant, Depo, or contraceptive pill, patch or ring] with consistent condom use;
  * Consistent condom use only
Participant report of adherence to DP strategy | 6 months
  By self-report from audio computer-assisted self-interviewing (ACASI) and telephone questionnaires; adherence is measured by three different outcomes:
  * Whether or not DP strategy was used at last sex
  * Whether or not DP strategy was used consistently during last 3 month time period
  * Estimated proportion of time adherent to DP strategy over last 3 months
Participant report of adherence to DP strategy | 9 months
  By self-report from audio computer-assisted self-interviewing (ACASI) and telephone questionnaires; adherence is measured by three different outcomes:
  * Whether or not DP strategy was used at last sex
  * Whether or not DP strategy was used consistently during last 3 month time period
  * Estimated proportion of time adherent to DP strategy over last 3 months
Participant report of adherence to DP strategy | 12 months
  By self-report from audio computer-assisted self-interviewing (ACASI) and telephone questionnaires; adherence is measured by three different outcomes:
  * Whether or not DP strategy was used at last sex
  * Whether or not DP strategy was used consistently during last 3 month time period
  * Estimated proportion of time adherent to DP strategy over last 3 months
Participant selection of an effective dual protection (DP) strategy | At enrollment visit
  Whether or not a participant self-reports having selected an effective DP strategy. An effective DP strategy is defined as one of the following:
  * Abstinence from vaginal sex;
  * Effective non-barrier contraceptive method [including intrauterine device (IUD), Implant, Depo, or contraceptive pill, patch or ring] with consistent condom use;
  * Consistent condom use only

SECONDARY OUTCOMES:
Participant level of reproductive health knowledge (percentage correct of knowledge questions) | 6 months
  Knowledge about contraceptives and STIs, as measured by correct answers to knowledge questions on ACASI questionnaires.
Participant intention to use DP strategy | 6 months
  Whether or not participant self-reports intention to use an effective DP strategy in the future, as measured by responses on ACASI questionnaires.
Participant reproductive health self-efficacy | 6 months
  Whether or not participant reported high self-efficacy for condom use, contraceptive use, and communication with partner on reproductive health topics, as measured by responses on ACASI questionnaires.
Participant report of STI testing | 6 months
  Frequency of self-reported STI testing by participant and partner(s) and result-sharing with partner(s), as measured by responses to ACASI questionnaires.
Participant report of partner communication | 6 months
  Self-reported frequency of communication with partner on reproductive health topics, as measured by responses on ACASI questionnaires.
Participant level of reproductive health knowledge (percentage correct of knowledge questions) | 12 months
  Knowledge about contraceptives and STIs, as measured by correct answers to knowledge questions on ACASI questionnaires.
Participant intention to use DP strategy | 12 months
  Whether or not participant self-reports intention to use an effective DP strategy in the future, as measured by responses on ACASI questionnaires.
Participant report of STI testing | 12 months
  Frequency of self-reported STI testing by participant and partner(s) and result-sharing with partner(s), as measured by responses to ACASI questionnaires.
Participant reproductive health self-efficacy | 12 months
  Whether or not participant reported high self-efficacy for condom use, contraceptive use, and communication with partner on reproductive health topics, as measured by responses on ACASI questionnaires.
Participant report of partner communication | 12 months
  Self-reported frequency of communication with partner on reproductive health topics, as measured by responses on ACASI questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Kottke, MD MPH MBA, Principal Investigator — Emory University; Grady Health System; Jessica Sales, PhD, Principal Investigator — Emory University; Athena Kourtis, MD PhD MPH, Principal Investigator — Centers for Disease Control and Prevention; Peggy Goedken, MPH, Study Director — Emory University
Locations (1):
- Grady Health System Teen Services Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kottke MJ, Sales JM, Goedken P, Brown JL, Hatfield-Timajchy K, Koumans EH, Hardin JW, Kraft JM, Kourtis AP. 2gether: A Clinic-Based Intervention to Increase Dual Protection from Sexually Transmitted Infections and Pregnancy in Young African American Females. J Womens Health (Larchmt). 2023 Jan;32(1):29-38. doi: 10.1089/jwh.2022.0209. Epub 2022 Nov 22. PMID 36413049
- [Derived] Kraft JM, Snead MC, Brown JL, Sales JM, Kottke MJ, Hatfield-Timajchy K, Goedken P. Reproductive Coercion Among African American Female Adolescents: Associations with Contraception and Sexually Transmitted Diseases. J Womens Health (Larchmt). 2021 Mar;30(3):429-437. doi: 10.1089/jwh.2019.8236. Epub 2020 Jul 13. PMID 32667837